CLINICAL TRIAL: NCT06862063
Title: Next Generation Sequencing (NGS) Analysis of Patients with Spontaneous Dissection of Cervical Arteries (sCeAD), a Multi-centric, Interventional, Cohort Study
Brief Title: Next Generation Sequencing Analysis of Patients with Spontaneous Dissection of Cervical Arteries
Acronym: NASCeAD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Collaborators: Fondazione Mondino (Other); University of Rome Tor Vergata (Other); Azienda Policlinico Umberto I (Other); San Camillo Hospital, Rome (Other); I.R.C.C.S. Fondazione Santa Lucia (Other); Fondazione I.R.C.C.S. Istituto Neurologico Carlo Besta (Other); Ospedale Policlinico San Martino (Other); Istituto Neurologico Mediterraneo Neuromed S. R. L (Other); IRCCS Istituto delle Scienze Neurologiche di Bologna (Other); Ospedale Guzzardi di Vittoria (Unknown); Santo Spirito Hospital, Italy (Other); Azienda Ospedaliera di Rilievo Nazionale A.Cardarelli (Other); Istituto Clinico Humanitas (Other); Ospedale V. Fazzi (Other)
Responsible Party: Principal Investigator, Frisullo Giovanni, Principal Investigator, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 6813
Record Dates: First submitted 2024-11-14; First posted 2025-03-06 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2024-11

CONDITIONS: Dissection Carotid Artery; Dissection Arterial; Dissecting Aneurysm
MeSH Terms: conditions — Aortic Dissection | interventions — Genetic Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Adult patients with spontaneous dissections of the Cervical arteries (Experimental)
  Interventions: Diagnostic Test: Genetic testing

INTERVENTIONS:
Diagnostic Test: Genetic testing — Each eligible patient will undergo a blood sample to perform a genetic analysis through Next Generation Sequencing (NGS) technique in order to analyze a high number of genes involved in the structure/function of connective tissue
  Other Names: Next generation sequencing analysis of an extended panel of genes

SUMMARY:
The goal of this observational study is to analyze the existence of a genetic predisposition in patients with spontaneous dissections of the cervical arteries (SCeAD).

The main questions it aims to answer are:

1. Which is the prevalence of pathogenic variants in genes coding for proteins involved in the structure or function of the connective tissue in adult patients with spontaneous dissections of the cervical arteries?
2. Which are the clinical characteristics of each single genetic variant identified?
3. Which are the clinical, radiological, laboratory variables associated with the finding of a pathogenic variant?
4. Are there differences between patients with SCeAD who have a pathogenic variant in a gene coding for proteins involved in the structure or function of the connective tissue and those who not?
5. There are differences in the risk of SCeAD recurrence between patients with SCeAD who have a pathogenic variant in a gene coding for proteins involved in the structure or function of the connective tissue and those who not?
6. There are differences in the risk of SCeAD recurrence based on the specific typology of genetic variant found?

Participants will be asked to undergo:

* a whole-CT total-body with contrast;
* a dysmorphological visit;
* a blood sampling for genetic testing;
* a neurological visit;
* Some follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

* Adult age (≥18 years);
* Presence of a dissection of one or more cervical arteries (carotid or vertebrobasilar district), defined as the finding, on an appropriate radiological examination (CT and/or MRI of the neck and brain district with/without contrast medium and/or digital subtraction angiography and/or echocolordoppler of the epiaortic vessels) of "intramural hematoma, pseudoaneurysmal dilation, intimal flap, double lumen, long tapering stenosis or occlusion ≥2 cm above the carotid bifurcation with finding of an aneurysmal dilation or a long tapering stenosis after recanalization of the vessel";
* At least one or more of the following criteria:

  * Radiological evidence on CT and/or MRI with/without contrast and/or digital subtraction angiography and/or color Doppler ultrasound of vessel wall anomalies (such as aneurysms, dissections, tortuosity, ectasia or vascular stenosis) in one or more vascular districts in addition to that of the known dissection;
  * Family history of:

    * vessel dissections and/or sudden death and/or cerebrovascular or cardiovascular diseases at a young age;
    * spontaneous perforation of internal organs and/or dehiscence and/or laxity of connective tissue (spontaneous prolapses);
  * dysmorphological abnormalities at the clinical examination (including Beighton score ≥5 or Marfan score ≥7), laboratory and/or radiological findings suggestive of connective tissue disease or other genetic condition known to be associated with the development of aneurysms or alterations of the vessel wall;
* Written informed consent

Exclusion Criteria:

* Recent history of trauma clearly related in type, location and dynamics to the development of dissection;
* Iatrogenic dissection following endovascular procedure;
* Exclusively intracranial dissection;
* Fibromuscular dysplasia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2030-12-01 (Estimated); Study Completion 2030-12-01 (Estimated)

PRIMARY OUTCOMES:
Definition of the percentage prevalence (n - %) of pathogenic variants in patients with Spontaneous Cervical Artery Dissection (SCeAD) | Through study completion, an average of 2 years and six months
  To define the percentage prevalence (n - %) of pathogenic variants of genes encoding proteins involved in the structure/function of connective tissue in patients with spontaneous dissection of the cervical arteries

SECONDARY OUTCOMES:
Evaluation of the percentage prevalence (n - %) of each pathogenic variant in genes encoding connective tissue proteins in patients with spontaneous dissection of the cervical arteries | Through study completion, an average of 2 years and six months
  Description of the typology and percentage prevalence (n - %) of individual pathogenic variants of genes encoding proteins involved in the structure/function of connective tissue in patients with spontaneous dissections of the Cervical arteries
Identification of clinical predictors of pathogenic variants in genes encoding connective tissue proteins in patients with spontaneous cervical artery dissection | Through study completion, an average of 2 years and six months
  Percentage prevalence (n - %) of clinical predictors of pathogenic variants in genes encoding proteins involved in the structure/function of connective tissue in patients with spontaneous dissection of the cervical arteries through multivariable regression models. In particular, clinical (eg. Beighton score, Marfan score, symptoms that lead to the finding of the dissection, etc), radiological (eg. the presence of vascular abnormalities in other vascular districts, the aspect of the cervical artery dissection at the US, CT, or MRI examination, etc.), and laboratory parameters (eg. hyperhomocisteinemia, immunological screening, CRP, etc.) will be compared between patients with spontaneous dissections of the cervical arteries who have a pthogenic variant of genes encoding for connective tissue proteins and those who not.
Assessment of the risk of artery dissection recurrence in patients with spontaneous cervical artery dissection carrying a pathogenic variant in those without through the ODD ratio | Through study completion, an average of 2 years and six months
  Comparison of the risk of recurrence of vascular dissections in the cervical arteries or in other vascular districts in patients with spontaneous cervical artery dissection carrying a pathogenic variant in genes encoding proteins involved in connective tissue structure/function and in those without it by calculating the ODD ratio
Definition of the prevalence of pathogenic variants in other genes | Through study completion, an average of 2 years and six months
  Percentage prevalence (n - %) of individual pathogenic variants of genes encoding proteins not involved in the structure/function of connective tissue in patients with spontaneous dissection of the cervical arteries and correlation of the same with individual clinical phenotypes;

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, Rome, Lazio, Italy

IPD SHARING:
Plan to Share IPD: No
There are not plans to make IPD available to other researchers as we will be dealing with highly sensitive data, such as genetic data.